CLINICAL TRIAL: NCT05565183
Title: Combined Study of ATrial Strain and Voltage by High Density Mapping in Young Patients With Atrial Fibrillation.
Acronym: CATS-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP190631
Record Dates: First submitted 2022-08-08; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-08

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Catheter Ablation; Atrial Cardiomyopathy
Keywords: Atrial Fibrillation; Atrial strain; High density electrical mapping; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diagnosed Atrial fibrillation and an indication of catheter ablation (Experimental)
  Interventions: Diagnostic Test: MRI (with injection of contrast product)

INTERVENTIONS:
Diagnostic Test: MRI (with injection of contrast product) — All patients included in the study will undergo two MRI examinations (with injection of contrast product) before and after the ablation procedure.

SUMMARY:
Atrial The treatment of atrial fibrillation (AF) includes 2 axes: the prevention of the cardio-embolic risk and rhythm control. The possibilities for this control are antiarrhythmic drugs and, above all, catheter ablation, an interventional cardiology technique which consists in treating the areas responsible for the initiation and perpetuation of AF by applying radiofrequency energy or cryotherapy to the myocardial tissue.

Limited research has been done on the combination of different parameters to manage AF, especially during the initial stage of the disease. A translational and multimodal approach could make it possible to better characterize this pathology and thus, help to adjust the therapeutic management for the patients.

The combined analysis of regional electrophysiological, morphological, and functional parameters of the left atrium could make it possible to better detect early atrial cardiomyopathy and predict recurrences of atrial fibrillation.

DETAILED DESCRIPTION:
The electrophysiological substrate for patients with persistent atrial fibrillation is heterogeneous with areas of atrial myocardium of low voltage amplitudes and areas of rapid fragmented signals in arrhythmia. The targets of ablation treatment in these cases are currently poorly defined. Several promising strategies have emerged, such as the isolation of fibrotic areas, low voltage.

An integration analysis of regional electrophysiological, morphological, and functional parameters of the left atrium, therefore, open up a new area of research that has not been studied to date and could help to better guide the therapeutic management of patients with AF.

The study aims to assess the association between regional and global myocardial strain abnormalities on magnetic resonance imaging (MRI) and the amplitude of the atrial intracardiac electrical potential, in young subjects with symptomatic AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 to 60 years
2. Established diagnosis of paroxysmal or persistent symptomatic atrial fibrillation (AF) for at least 3 months with indication of catheter ablation
3. AF episode documented by ECG in the last 12 months
4. Structurally healthy heart, with an LVEF> 50%, an interventricular septum <12 mm and an OG volume <40mL / m ² by TTE
5. Having given their informed consent in writing
6. Affiliated with or entitled to a French social security scheme

Exclusion Criteria:

1. Mitral valve disease with grade 2 to 4 insufficiency
2. Heart failure (NYHA stage II to IV in sinus rhythm and LVEF < 50%), hypertrophic heart disease or congenital heart disease
3. Contraindication to oral anticoagulation
4. Intracardiac thrombus
5. History of ablation of the left atrium
6. History of heart surgery
7. Contraindication to performing MRI or using the DOTAREM™ contrast medium (pacemaker, defibrillator, prosthesis, old generation heart valves, old generation ferromagnetic vascular surgical clips, treatment type endocranial aneurysms, neurosimulator, cochlear implants, automated injection device such as insulin pump, and more generally any non-removable electronic medical device or equipment, kidney disease with GFR < 30 mL/min, hypersensitivity to gadoteric acid or to excipients)
8. History of myocardial infarction or coronary angioplasty within the last three months
9. Chronic obstructive pulmonary disease
10. Under guardianship or curatorship
11. Women who are pregnant, breastfeeding or of childbearing age in the absence of effective contraception
12. Participation in another interventional research involving a health product

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between the regional and global longitudinal strain peaks (percent (%)) and voltage (millivoltage(mV)) of the left atrium measured by MRI and catheter ablation | 1 month

SECONDARY OUTCOMES:
Localization in the left atrium and area of low amplitude electrogram areas (<0.5 mV, <0.3 mV and <0.1 mV) measured during the ablation procedure | 1 month
Localization in the left atrium and areas of fragmented atrial complexes measured during the ablation procedure | 1 months
Local atrial impedance measured by ablation catheter | 1 months
Contact force measured by ablation catheter | 1 month
Local impedance drop measured during radiofrequency delivery | 1 month
Duration of the ablation for each radiofrequency delivery | 1 month
Localization of the segmental and regional alteration of the myocardium in the left atrium measured during MRI | 3 months
Localization of zones with impaired 4D flow in the left atrium measured during MRI | 3 months
Left atrium volume (milliliter (mL)) measured during MRI | 3 months
Localization of areas of late enhancement in the left atrium | 3 months
Lesion transmurality performed by ablation in each segment of the pulmonary veins | 3 months
Subcutaneous measurement (AGE Reader) which combines aging and accumulation of glycated proteins in the subcutaneous tissue measured during MRI | 3 months
Volumes (milliliter (ml)) of the left atrium: in the basal state and after passive filling measured during echocardiography | 1 month
Analysis of the longitudinal deformation (strain) in speckle tracking in the basal state and after passive measured during echocardiography | 1 month
Absence of atrial fibrillation occurrence | 12 months
Absence of persistent atrial fibrillation occurrence | 12 months
Absence of atrial tachycardia or atrial flutter occurrence after catheter ablation | 12 months
Absence of palpitation occurrence after catheter ablation | 12 months
6-minute walking test to assess exercise capacity | 1 month
Differences in the volumes (milliliter (ml)) of the left atrium (maximum, minimum, atrial pre-systole) between the segmentation performed manually and the segmentation obtained by learning transfer | 3 months
Distance between areas of low voltages identified by the cartography and areas of late 3D enhancement identified by MRI, measurement based on the volume (milliliter (ml)) resulting from CT-scan and MRI fusion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BADENCO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut de Cardiologie de la Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal